CLINICAL TRIAL: NCT04304092
Title: Addressing Individual Variability in Response to Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID associated costs have reduced the available budget , and the ability to recruit participants from the community. These two factors combined do not allow us to perform the trial as originally planned.
Sponsor: Dr. Robert Ross (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Robert Ross, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ross2019
Record Dates: First submitted 2020-02-28; First posted 2020-03-11 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2021-09

CONDITIONS: Exercise; Cardiorespiratory Fitness
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Masking Description: exercise trial, no blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low amount, low intensity (Experimental)
  Interventions: Other: Exercise
- Low amount, high intensity (Experimental)
  Interventions: Other: Exercise
- High Amount, low intensity (Experimental)
  Interventions: Other: Exercise
- High Amount, high intensity (Experimental)
  Interventions: Other: Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise — Participants will exercise under supervision. Exercise dose will vary by amount and intensity
  Arms: High Amount, high intensity; High Amount, low intensity; Low amount, high intensity; Low amount, low intensity

SUMMARY:
In this proposal, the investigators challenge the assumption that following the physical activity guidelines implies benefit for ALL adults, and that if benefit is not achieved in response to first line therapy, it will be by simply exercising more. Thus, for improving cardiorespiratory fitness and cardiometabolic risk factors, unanswered questions include: 1) To what extent, regardless of exercise amount or intensity, is exercise not associated with benefit? Demonstration of a resistance to benefit through exercise in a substantial number of adults would be a novel and important finding, would counter the assumptions of many if not most health care practitioners, and could have immediate and direct application in all health care settings. 2) To what extent will non-responders to first line therapy (150 min/wk) be required to increase exercise amount or intensity to achieve benefit? 3) To what extent will failure to improve CRF segregate (be associate with) with cardiometabolic risk factors? The investigators propose that adults who remain exercise resistant for improvement in CRF and cardiometabolic risk despite increasing amount or intensity are at high risk of metabolic disease and consequently, are candidates for alternative treatment strategies. 4) To what extent is biological sex and/or phenotype a determinant of response or non-response to exercise?

DETAILED DESCRIPTION:
The trial has three objectives:

Primary objective: Determine whether alterations in exercise amount and intensity improves the rate of clinically meaningful improvements in aerobic exercise capacity as measured by cardiorespiratory fitness (CRF, VO2peak) among adults.

Secondary objective: Determine whether common cardiometabolic risk factors segregate with respect to variation in CRF to first line therapy in adults, and, whether clinically meaningful improvements in cardiometabolic risk factors segregate with associated improvement in CRF.

Tertiary objective: Identify whether biological sex and/or phenotype are determinants of variation in CRF and cardiometabolic risk factors in response to first line therapy, and, whether they predict variability in CRF response to alterations in exercise dose.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle (planned physical activity for one day per week or less).
* Weight stable (± 2 kg) for 6 months prior to the beginning of the study.
* BMI between 20 and 40 kg/m2.

Exclusion Criteria:

* Physical impairment which would make the intervention very difficult or unsafe according to doctor's advice.
* Diabetes, current smokers.
* Plan to move from the area in next 8 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Measured at baseline and every 4 weeks for 32 weeks.
  Cardiorespiratory fitness will be determined using direct (open circuit spirometry) measures of oxygen consumption (expressed in L/min) obtained during a maximal treadmill test.

SECONDARY OUTCOMES:
Change in cardiometabolic risk factors | Measured at baseline, 16 and 32 weeks.
  Fasting glucose (mmol/L)
Change in cardiometabolic risk factors | Measured at baseline, 16 and 32 weeks.
  Fasting LDL- and HDL-cholesterol (mmol/L)
Change in cardiometabolic risk factors | Measured at baseline, 16 and 32 weeks.
  fasting insulin (pmol/L)
Change in cardiometabolic risk factor | Measured at baseline, 16 and 32 weeks.
  fasting triglycerides (mmol/L)